CLINICAL TRIAL: NCT07215312
Title: A Phase 2, Randomized, Open-Label, Comparator-Controlled Trial to Evaluate the Efficacy and Safety of LY3938577 in Study Participants, With Type 2 Diabetes Previously Treated With Basal Insulin
Brief Title: A Study of LY3938577 in Participants With Type 2 Diabetes Previously Treated With Basal Insulin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27409; J4P-MC-IYAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-09; First posted 2025-10-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycemic control; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Hyperglycemia | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3938577 (Experimental): Participants will receive LY3938577 subcutaneously (SC)
  Interventions: Drug: LY3938577
- Degludec (Active Comparator): Participants will receive degludec SC
  Interventions: Drug: Degludec

INTERVENTIONS:
Drug: LY3938577 — Administered SC
  Arms: LY3938577
Drug: Degludec — Administered SC
  Arms: Degludec

SUMMARY:
The purpose of this study is to see how well LY3938577 works and how safe it is compared to degludec in people with type 2 diabetes. Participation in the study will last about 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Are receiving ≥20 units of basal insulin per day and ≤55 units/day and ≤1.5 units/kg/day at screening
* Have hemoglobin A1c (HbA1c) 7.5% to 10.5% inclusive
* Have a body mass index (BMI) of 20 or higher and less than 35 kilograms per square meter (kg/m2)

Exclusion Criteria:

* Have type 1 diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Glucose Time in Range Between 70 and 180 mg/dL Inclusive (Non-Inferiority Analysis) | Baseline through Week 20

SECONDARY OUTCOMES:
Change from Baseline in Glucose Time in Range Between 70 and 180 mg/dL Inclusive (Superiority Analysis) | Baseline through Week 20
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 20
Pharmacokinetics (PK): Average Concentration of LY3938577 | Baseline through Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (20):
  - Tucson Clinical Research Institute, Tucson, Arizona
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - Encore Medical Research, Hollywood, Florida
  - Clinical Research of Central Florida, Lakeland, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Accellacare - Wilmington, Wilmington, North Carolina
  - AMR Clinical, Norman, Oklahoma
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Chrysalis Clinical Research, St. George, Utah
- Argentina (6):
  - CIPREC, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Instituto Centenario, CABA
  - Instituto Médico Catamarca IMEC, Rosario

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3938577 in Participants With Type 2 Diabetes Previously Treated With Basal Insulin — https://trials.lilly.com/en-US/trial/659897